CLINICAL TRIAL: NCT00473889
Title: A Phase II/III Randomized, Double-Blind Study of Paclitaxel Plus Carboplatin in Combination With Vorinostat or Placebo in Patients With Stage IIIB (With Pleural Effusion) or Stage IV Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: A Clinical Trial of Vorinostat (MK0683, SAHA) in Combination With FDA Approved Cancer Drugs in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)(0683-056)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated based on the recommendation by the DSMB following a pre-planned protocol interim analysis because the endpoint was not achieved.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0683-056; MK0683-056; 2006_539
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Results first posted 2009-10-12 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Stage IIIB or IV Non-Small Cell Lung Cancer
MeSH Terms: interventions — Vorinostat; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): vorinostat; IV paclitaxel; IV carboplatin
  Interventions: Drug: vorinostat; Drug: Comparator: paclitaxel; Drug: Comparator: carboplatin
- 2 (Placebo Comparator): Placebo; IV paclitaxel; IV carboplatin
  Interventions: Drug: Comparator: paclitaxel; Drug: Comparator: carboplatin; Drug: Comparator: placebo

INTERVENTIONS:
Drug: vorinostat — vorinostat 400 mg capsules once daily. Up to 6 months of treatment
  Other Names: Zolinza
  Arms: 1
Drug: Comparator: paclitaxel — intravenous (IV) paclitaxel 200 mg/m2. Up to 6 months of treatment
  Other Names: Taxol
Drug: Comparator: carboplatin — intravenous (IV) carboplatin AUC 6mg/min/ml. Up to 6 months of treatment.
  Other Names: Paraplatin
Drug: Comparator: placebo — vorinostat 400 mg placebo capsules once daily. Up to 6 months of treatment
  Arms: 2

SUMMARY:
This Phase III clinical trial which incorporates an initial Phase II component will determine the survival of advanced Non-small cell lung cancer patients when treated with MK0683 and paclitaxel plus carboplatin

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age who have confirmed diagnosis of Non-small Cell Lung Cancer
* Patients with no systemic prior systemic treatment for lung cancer except patients at least 12 months from prior adjuvant therapy
* Adequate bone marrow,kidney and liver function
* Must be recovered and at least 4 weeks from major surgery or radiation
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
* Men and women must agree to use birth control during the study
* Women able to have children must have a negative pregnancy test 14 days before study enrollment

Exclusion Criteria:

* Patients with prior treatment with other investigational agents less than 4 weeks before study enrollment
* Pregnant or nursing female patients
* Patients who are HIV positive
* Patients who have Hepatitis A, B, or C
* Patients unable to take study medication by mouth
* Patients with untreated brain cancer
* Patient eligible for treatment with bevacizumab and for whom bevacizumab is available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Beaumont H, Souchet S, Labatte JM, Iannessi A, Tolcher AW. Changes of lung tumour volume on CT - prediction of the reliability of assessments. Cancer Imaging. 2015 Oct 31;15:17. doi: 10.1186/s40644-015-0052-2. PMID 26521238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 99 investigative sites worldwide. The first patient's first visit was 16 May 07 and the last patient's last visit was 12 Dec 2008.
Pre-assignment Details: Randomized participants were stratified by Stage (IIIB versus IV), geographic region and eligibility for treatment with bevacizumab prior to treatment assignment.
Groups:
- Vorinostat + Paclitaxel + Carboplatin: Experimental arm: Vorinostat capsules (400 mg) once daily on Days -4 through 10 of Cycle 1 (25 day treatment cycle) and Days 1 through 14 of each subsequent 21 day treatment cycle; paclitaxel (200 mg/m2) and carboplatin (area under concentration/time curve of 6 mg/min/mL) administered by intravenous (IV) infusion on Day 1 of each treatment cycle.
- Placebo + Paclitaxel + Carboplatin: Placebo Comparator arm: Placebo capsules once daily on Days -4 through 10 of Cycle 1 (25 day treatment cycle) and Days 1 through 14 of each subsequent 21 day treatment cycle; paclitaxel (200 mg/m2) and carboplatin (area under concentration/time curve of 6 mg/min/mL) administered by intravenous (IV) infusion on Day 1 of each treatment cycle.
Period: Overall Study
Arm/Group | Vorinostat + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Started | 126 | 127
Completed | 43 | 63
Not Completed | 83 | 64
Not completed — Did not receive study medication | 1 | 4
Not completed — Adverse Event | 30 | 17
Not completed — Protocol Violation | 4 | 2
Not completed — Lack of Efficacy | 28 | 29
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 10 | 5
Not completed — Trial Terminated | 3 | 6
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 126 | 127 | 253
Age, Customized [Number; unit: participants]
  Less Than 65 years | 70 | 89 | 159
  65 years or Older | 56 | 38 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 56 | 90
  Male | 92 | 71 | 163
Race/Ethnicity, Customized [Number; unit: participants]
  White | 79 | 79 | 158
  Black | 3 | 4 | 7
  Asian | 31 | 32 | 63
  American Indian or Alaskan Native mix | 13 | 12 | 25
Cancer Stage [Number; unit: Participants]
  IIIB | 14 | 15 | 29
  IV | 112 | 112 | 224
Eligibility to receive treatment with Bevacizumab [Number; unit: Participants]
  Eligible | 70 | 63 | 133
  Ineligible | 55 | 60 | 115
  Unknown | 1 | 4 | 5
Geographic region where the participant lived [Number; unit: Participants]
  North America | 25 | 27 | 52
  Europe (United Kingdom, Italy, Germany, and Spain) | 41 | 40 | 81
  Asia | 22 | 24 | 46
  Rest of the World | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Defined as the time from date of randomization to death due to any cause. Patients without documented death at the time of the final analysis will be censored at the date of the last follow-up.
Time Frame: Start of treatment to death
Population: Intention-to-treat (ITT) population is defined as all randomized participants. Participants are counted in the group to which they are randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Vorinostat + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 126 | 127
Months | 11.0 [0.2 to 17.3] | 14.0 [0.03 to 18.7]
Statistical Analysis 1: Comparison: Placebo + Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.992, Stratified Log Rank — This is a one sided p-value, which corresponds to the null hypothesis; Disease stage and bevacizumab eligibility are the stratification factors in the stratified log rank test

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in sum of the longest diameter of all target lesions, the appearance of a new lesion, or an increase in non-target lesions.
Time Frame: Start of treatment to disease progression or death
Population: Full analysis set
  (FAS) population defined as all randomized participants who have received at least one dose of study medication. There are 253 participants randomized in the study 5 didn't take any study medication. Therefore, 248 participants are included in this analysis population.
Measure: Median (Full Range); unit: Months
Arm/Group | Vorinostat + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 125 | 123
Months | 4.3 [0.03 to 13.4] | 5.5 [0.03 to 13.8]
Statistical Analysis 1: Comparison: Placebo + Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.862, Finkelstein's Interval Censored Method — This is a one sided p-value, which corresponds to the null hypothesis; Disease stage and bevacizumab eligibility are the stratification factors in the Finkelstein's Interval Censored Method Model

3. Secondary Outcome: Number of Participants Who Had a Disease Response to Treatment
Description: Response to treatment is defined as a complete response (CR) or partial response (PR) to treatment. Confirmation of response required a second assessment performed at least 4 weeks after the initial assessment. (PR is defined as at least a 30% reduction in sum of the longest diameter of all target lesions and no increase in non-target lesions).
Time Frame: Every 42 days from start of treatment until disease response
Population: Full analysis set
  (FAS) population is defined as all randomized participants who have received at least one dose of study medication. There are 253 participants randomized in the study. Five (5) didn't take any study medication. Therefore, 248 participants are included in this analysis population.
Measure: Number; unit: Participants
Arm/Group | Vorinostat + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Number analyzed (Participants) | 125 | 123
Participants
  Responder | 28 | 36
  Non-Responder | 97 | 87
Statistical Analysis 1: Comparison: Placebo + Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.899, Stratified Miettinen and Nurminen — This is a one sided p-value, which corresponds to the null hypothesis; Disease stage and bevacizumab eligibility are the stratification factors in the stratified Miettinen and Nurmimen method

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time the patient signed the informed consent form until 30 days after the last dose of study medications. Serious Adverse Events were followed until resolution.
Description: The 5 untreated patients on study are not counted in the Adverse Events tables. Further, one patient was randomized to vorinostat but took placebo; and one patient, randomized to placebo, started vorinostat for 4 days before using placebo. Both patients are counted in the placebo group for Adverse Events, yielding 124 patients in each group.
Arm/Group | Vorinostat + Paclitaxel + Carboplatin | Placebo + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 63/124 | 45/124
Other Adverse Events (participants affected / at risk) | 114/124 | 117/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat + Paclitaxel + Carboplatin (N=124) | Placebo + Paclitaxel + Carboplatin (N=124)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 5
Neutropenia (Blood and lymphatic system disorders) | 9 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 6 | 1
Death (General disorders) | 2 | 1
Fatigue (General disorders) | 3 | 1
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 9
Pulmonary sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 2 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 11
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat + Paclitaxel + Carboplatin (N=124) | Placebo + Paclitaxel + Carboplatin (N=124)
Anaemia (Blood and lymphatic system disorders) | 51 | 42
Leukopenia (Blood and lymphatic system disorders) | 13 | 18
Lymphopenia (Blood and lymphatic system disorders) | 9 | 10
Neutropenia (Blood and lymphatic system disorders) | 53 | 55
Thrombocytopenia (Blood and lymphatic system disorders) | 45 | 23
Tinnitus (Ear and labyrinth disorders) | 0 | 5
Vision blurred (Eye disorders) | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6
Constipation (Gastrointestinal disorders) | 34 | 26
Diarrhoea (Gastrointestinal disorders) | 43 | 36
Dry mouth (Gastrointestinal disorders) | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 8 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 4
Gastritis (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 46 | 39
Stomatitis (Gastrointestinal disorders) | 12 | 11
Vomiting (Gastrointestinal disorders) | 34 | 24
Asthenia (General disorders) | 27 | 18
Chills (General disorders) | 5 | 4
Fatigue (General disorders) | 28 | 32
Oedema peripheral (General disorders) | 11 | 13
Pyrexia (General disorders) | 21 | 11
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 0
Influenza (Infections and infestations) | 0 | 5
Pneumonia (Infections and infestations) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 12
Urinary tract infection (Infections and infestations) | 7 | 5
Alanine aminotransferase increased (Investigations) | 10 | 13
Aspartate aminotransferase increased (Investigations) | 9 | 9
Blood alkaline phosphatase increased (Investigations) | 9 | 7
Weight decreased (Investigations) | 6 | 10
Anorexia (Metabolism and nutrition disorders) | 34 | 31
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 9
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 13
Dizziness (Nervous system disorders) | 9 | 12
Dysgeusia (Nervous system disorders) | 11 | 9
Headache (Nervous system disorders) | 13 | 12
Lethargy (Nervous system disorders) | 4 | 1
Peripheral motor neuropathy (Nervous system disorders) | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 51 | 61
Tremor (Nervous system disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 6 | 7
Insomnia (Psychiatric disorders) | 19 | 15
Dysuria (Renal and urinary disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 41 | 47
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 10
Rash (Skin and subcutaneous tissue disorders) | 18 | 13
Deep vein thrombosis (Vascular disorders) | 4 | 0
Hypertension (Vascular disorders) | 4 | 5
Hypotension (Vascular disorders) | 1 | 4
Thrombophlebitis superficial (Vascular disorders) | 4 | 2

LIMITATIONS AND CAVEATS:
The study was stopped following a pre-planned interim analysis because the goal for this study to continue was not met, based on 100 events, a reduction in the hazard ratio for progression-free survival by > 23% with a one-sided p-value < 0.1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.